CLINICAL TRIAL: NCT05312775
Title: Single Versus Double-layer Closure of The Cesarean Scar In Niche Development: A Randomized Clinical Trial
Brief Title: Niche In CEsarean Scar Trial (NICEST)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Thi Thu Ha (Other)
Responsible Party: Sponsor-Investigator, Nguyen Thi Thu Ha, Deputy Director, Hanoi Obstetrics and Gynecology Hospital
Organization: Hanoi Obstetrics and Gynecology Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PSHN.0005.2021
Record Dates: First submitted 2022-03-01; First posted 2022-04-06 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Niche
Keywords: single-layer uterine closure; double-layer uterine closure; niche

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-layer uterine closure (Active Comparator): Women will undergo a CD following a standard way with respect to the mode of hysterotomy, non-closure of the peritoneum. The control group will receive a single-layer closure using unlocked continuous running multifilament sutures and the endometrial layer will be included
  Interventions: Procedure: Single-layer uterine closure
- Double-layer uterine closure (Active Comparator): Women will undergo a CD following a standard way with respect to the mode of hysterotomy, non-closure of the peritoneum. In the intervention group, double-layer closure of the uterus will be performed using unlocked multifilament continuous running sutures for both layers and the endometrial layer will be included in the first layer. The second layer is a continuous running suture that imbricates the first layer
  Interventions: Procedure: Double-layer uterine closure

INTERVENTIONS:
Procedure: Double-layer uterine closure — In the intervention group, double-layer closure of the uterus will be performed using unlocked multifilament continuous running sutures for both layers and the endometrial layer will be included in the first layer. The second layer is a continuous running suture that imbricates the first layer
  Arms: Double-layer uterine closure
Procedure: Single-layer uterine closure — The control group will receive a single-layer closure using unlocked continuous running multifilament sutures and the endometrial layer will be included
  Arms: Single-layer uterine closure

SUMMARY:
Rationale: Cesarean delivery (CD) rates are increasing rapidly worldwide. The consequences of cesarean section not only affect the next pregnancies such as uterine rupture or malplacentation but also cause many gynecological complications or infertility due to the formation of cesarean scar defect (CSD) or Niche. One of the major factors for Niche formation is the techniques of hysterotomy closure at the time of cesarean delivery. Most common hysterotomy closures include single and double layers closure. However, there is limited literature to prove which technique decreases niche creation and associated gynecological complications.

Objective: To compare the effect of uterine closure techniques during CD on the formation of Niche evaluated on transvaginal ultrasound and gynecological complications.

Study design: a double-blinded, single-center, randomized clinical trial. Setting: Hanoi Obstetrics & Gynecology Hospital (HOGH), Viet Nam. Study population: All women at gestational age ≥ 37 0/7 weeks who undergo a primary CD (planned or unplanned).

Intervention: After informed consent, women will be randomized to either unlocked single layer closure or unlocked double-layer closures of cesarean uterine scar in a 1:1 ratio Primary outcome: The proportion of Niche over time (at 6, 12, 18, 24 months after CD) in the two groups.

Power calculation: A sample size of 389 women is needed for each group. Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: Both uterine closure methods followed by the Vietnam Ministry of Health (VN-MOH), transvaginal ultrasound is also not harmful. It is believed that there are no potential increased risks to patients taking part in this trial because of the standard care and management they receive.

DETAILED DESCRIPTION:
Pregnancies at term, indicated for cesarean delivery for the first time, will be fully consulted information related to this study before surgery. Written consent will be obtained from each eligible pregnant woman before randomization into the study.

After signing the informed consent form, eligible women will be randomly assigned in a 1:1 ratio to receive either single-layer closure or double-layer closure, using block randomization with a variable block size of 4, 6. The computer-generated random list will be prepared by an independent statistician who has no other involvement in the study. To ensure allocation concealment, opaque and sealed envelopes will be prepared and controlled by two administrative staff in the Clinical Trial Unit who have no involvement in clinical work. Whenever there is an eligible participant, these two staff will hand over the envelope in sequence to the clinician. As the result, surgeons will not be blinded, but participants and sonographers will be unaware of closure techniques. Apart from randomization, patients will be followed up and treated according to local protocol.

The cesarean section with two uterine scar closure techniques will be performed by well-trained obstetricians. Participants and sonographers will be blinded for the closure technique.

Intervention (double-layer closure) In both study groups, women will undergo a CD following a standard way with respect to the mode of hysterotomy, non-closure of the peritoneum. In the intervention group, double-layer closure of the uterus will be performed using unlocked multifilament continuous running sutures for both layers and the endometrial layer will be included in the first layer. The second layer is a continuous running suture that imbricates the first layer.

Control group (single-layer closure) The control group will receive a single-layer closure using unlocked continuous running multifilament sutures and the endometrial layer will be included.

Complication during surgery

The cases that have complications during surgery will be excluded from the study. Complications encompass:

* Maternal mortality
* Maternal admitted ICU
* Hysterectomy
* Damage to internal organs (bowel, bladder or ureters).
* Complications during postoperative period requiring further surgery. Follow-up Participants will be contacted via telephone to notify about follow-up visits within 10 days of the first day of every menstrual cycle at 6 months, 12 months, 18 months, 24 months (give or take 2 weeks).

Every regular follow-up visit, the participants will be examined and transvaginal ultrasound followed by saline infusion sonohysterography to evaluate Niche. The ultrasound evaluation is standardized as proposed by the latest standard of ISUOG(2019).

Reproductive outcomes at two years follow-up: Percentage of women that conceived at any time during the follow-up duration, time of conception, and results of said pregnancies (ongoing pregnancy, terminated pregnancy due to medical/ social indication).

Niche evaluation Every regular follow-up visit, the participants will be examined and transvaginal ultrasound followed by sonohysterography to evaluate Niche. The Niche evaluation is standardized as proposed by the latest standard of ISUOG(2019).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who undergo a primary CD (planned or unplanned)
* Age ≥ 18 years.
* Gestational age ≥ 37 0/7 weeks

Exclusion Criteria:

* Previous major uterine surgery (e.g. laparoscopic or laparotomic fibroid resection, septum resection).
* Women with abnormal menstrual bleeding (e.g. cervical dysplasia, communicating hydrosalpinx, uterine anomaly or endocrine disorders disturbing ovulation, drugs, polyps, fibroids, etc.).
* Women with dysmenorrhea, dyspareunia, suprapubic pain.
* Abnormal placenta: Placenta privia, Placenta percreta… in the current pregnancy.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 938 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of Niche at 6 months after cesarean delivery of Single-layer uterine closure group | from delivery to 6 months from delivery
  The proportion of Niche at 6 months after cesarean delivery of Single-layer uterine closure group.
The proportion of Niche at 12 months after cesarean delivery of Single-layer uterine closure group | from delivery to 12 months from delivery
  The proportion of Niche at 12 months after cesarean delivery of Single-layer uterine closure group.
The proportion of Niche at 18 months after cesarean delivery of Single-layer uterine closure group | from delivery to 18 months from delivery
  The proportion of Niche at 18 months after cesarean delivery of Single-layer uterine closure group.
The proportion of Niche at 24 months after cesarean delivery of Single-layer uterine closure group | from delivery to 24 months from delivery
  The proportion of Niche at 24 months after cesarean delivery of Single-layer uterine closure group.
The proportion of Niche at 6 months after cesarean delivery of Double-layer uterine closure group | from delivery to 6 months from delivery)
  The proportion of Niche at 6 months after cesarean delivery of Double-layer uterine closure group.
The proportion of Niche at 12 months after cesarean delivery of Double-layer uterine closure group | from delivery to 12 months from delivery
  The proportion of Niche at 12 months after cesarean delivery of Double-layer uterine closure group.
The proportion of Niche at 18 months after cesarean delivery of Double-layer uterine closure group | from delivery to 18 months from delivery
  The proportion of Niche at 18 months after cesarean delivery of Double-layer uterine closure group.
The proportion of Niche at 24 months after cesarean delivery of Double-layer uterine closure group | from delivery to 24 months from delivery
  The proportion of Niche at 24 months after cesarean delivery of Double-layer uterine closure group.

SECONDARY OUTCOMES:
Number of participants with post-partum hemorrhage. | Within 24 hours from delivery
  Defined as blood loss more than 1000ml with 24 hours after cesarean delivery
Number of participants having uterine atony | During operation
  Defined as use of two or more uterotonics other oxytocin; other surgical interventions such as compression by hand and/or sutures, uterine arteries ligation, embolization, hypogastric arteries ligation, or balloon tamponade
Number of participants with maternal infection | from delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Maternal infection as defined:
  * Fever: defined as axillary temperature ≥ 37.5 degrees Celsius.
  * Start of intravenous broad-spectrum antibiotics (with evidence of infection confirmed by clinical and subclinical presentation)
  * Endometritis, myometritis or urinary tract infection (proven positive vaginal discharge/urine culture)
Number of participants having postmenstrual spotting in women with Niche | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Postmenstrual spotting is brownish discharge for more than two days at the end of menstruation with a total duration (menstruation and spotting) of more than seven days, or intermenstrual bleeding that starts after the end of menstruation, assessed at 6 months, 12 months, 18 months and 24 months after delivery.
Duration of postmenstrual spotting in women with Niche | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Duration of postmenstrual spotting in women with Niche defined as the average number of days of postmenstrual spotting in 6 months, in which duration of postmenstrual spotting in each month will be counted as follows: days with brownish discharge (more than two days) when the total duration of menstruation and spotting exceeds seven days plus days with intermenstrual bleeding, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery.
Number of participants suffering from dysmenorrhea in women with Niche | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Number of participants suffering from dysmenorrhea in women with Niche, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery
Dysmenorrhea severity in women with Niche | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Participants with dysmenorrhea self-assessed pain levels and scored 1 to 10 rely on the Numeric Rating Scale (NRS). The average score in span of 6 months will be calculated and the highest score will be noticed to reveal dysmenorrhea severity at 6 months, 12 months, 18 months, 24 months after cesarean delivery
Number of participants suffering from suprapubic pain in women with Niche | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Number of participants suffering from suprapubic pain in women with Niche, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery
Suprapubic pain severity in women with Niche | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Participants with suprapubic pain self-assessed pain levels and scored 1 to 10 rely on the Numeric Rating Scale (NRS). The average score in span of 6 months will be calculated and the highest score will be noticed to reveal suprapubic pain severity at 6 months, 12 months, 18 months, 24 months after cesarean delivery
Number of participants suffering from dyspareunia in women with Niche | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Number of participants suffering from dyspareunia in women with Niche, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery
Dyspareunia severity in women with Niche | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Participants with dyspareunia self-assessed pain levels and scored 1 to 10 rely on the Numeric Rating Scale (NRS). The average score in span of 6 months will be calculated and the highest score will be noticed to reveal dyspareunia severity at 6 months, 12 months, 18 months, 24 months after delivery
Niche length | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  The length at Niche base will be measured in the sagittal plane on transvaginal ultrasound, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery.
Niche depth | : from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  The largest depth of Niche will be measured in the sagittal plane on ultrasound, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery.
Number of branches of Niche | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Number of branches of Niche will be measured in the transverse plane on transvaginal ultrasound, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery.
Residual myometrial thickness (RMT) | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Thinnest point of residual myometrial thickness will be measured in the sagittal plane on transvaginal ultrasound, regardless of direction (measured perpendicular to serosa but not necessarily to uterine cavity), from the main Niche or branch with the thinnest RMT. Fibroid is not included in RMT measurement, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery.
Ratio of residual myometrial thickness per adjacent myometrial thickness (RMT/AMT) | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Adjacent myometrial thickness will be measured close to Niche in the sagittal plane on transvaginal ultrasound, where myometrium is thickness. Ratio of RMT/AMT will be assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery.
Niche-vesicovaginal fold distance | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Distance between Niche and vesicovaginal fold will be measured in the sagittal plane on transvaginal ultrasound, from level of top main Niche (where residual myometrial thickness is smallest (dotted line)) to vesicovaginal fold, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery.
Niche-external os distance | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Distance between niche and external os will be measured parallel to cervical canal, from most distal point of niche to external os in the sagittal plane on transvaginal ultrasound, assessed at 6 months, 12 months, 18 months and 24 months after cesarean delivery.
Evaluating the correlation between Niche characteristics and gynecological symptoms | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Correlation between characteristics of Niche (include length, depth, branches, RMT, RMT/AMT, Niche-vesicovaginal fold distance and Niche-external os distance) and gynecological symptoms (involve postmenstrual spotting, dysmenorrhea, suprapubic pain and dyspareunia) will be analyzed at 6 months, 12 months, 18 months and 24 months after cesarean delivery
Evaluating factors contributing to Niche development | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Correlation between Niche formation and risk factors include labor (cervical dilation, duration of labor), planned or unplanned cesarean section, maternal factors, short-term outcomes such as uterine atony, post-partum hemorrhage, post-partum blood transfusion, maternal infection will be analyzed at 6 months, 12 months, 18 months and 24 months after cesarean delivery
Comparison between the rate of niche detection by regular TVUS and sonohysterography | from delivery to 6 months, 12 months, 18 months, 24 months after cesarean delivery, up to 24 months from delivery
  Comparison between rate of niche detection (percentage) in all follow-up events by regular TVUS and sonohysterography

OTHER OUTCOMES:
Reproductive outcome during 2 years of follow-up | 24 months from delivery
  Percentage of women that conceived at any time during 2 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anh D Nguyen, PhD. MD, Study Director — Hanoi Obstetric and Gynecology Hospital; Yves Ville, PhD. MD, Study Chair — Hôpital Necker-Enfants Malades; Ha TT Nguyen, PhD.MD, Principal Investigator — Hanoi Obstetric and Gynecology Hospital; Giang TT Duong, MD, Principal Investigator — Hanoi Obstetric and Gynecology Hospital
Locations (1):
- Hanoi Obstetrics and Gynecology Hospital, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delport S. Global epidemiology of use of and disparities in caesarean sections. Lancet. 2019 Jul 6;394(10192):23-24. doi: 10.1016/S0140-6736(19)30717-2. Epub 2019 Jul 4. No abstract available. PMID 31282354
- [Background] Naji O, Wynants L, Smith A, Abdallah Y, Saso S, Stalder C, Van Huffel S, Ghaem-Maghami S, Van Calster B, Timmerman D, Bourne T. Does the presence of a Caesarean section scar affect implantation site and early pregnancy outcome in women attending an early pregnancy assessment unit? Hum Reprod. 2013 Jun;28(6):1489-96. doi: 10.1093/humrep/det110. Epub 2013 Apr 12. PMID 23585560
- [Background] Naji O, Wynants L, Smith A, Abdallah Y, Stalder C, Sayasneh A, McIndoe A, Ghaem-Maghami S, Van Huffel S, Van Calster B, Timmerman D, Bourne T. Predicting successful vaginal birth after Cesarean section using a model based on Cesarean scar features examined by transvaginal sonography. Ultrasound Obstet Gynecol. 2013 Jun;41(6):672-8. doi: 10.1002/uog.12423. PMID 23371440
- [Background] Roberge S, Demers S, Berghella V, Chaillet N, Moore L, Bujold E. Impact of single- vs double-layer closure on adverse outcomes and uterine scar defect: a systematic review and metaanalysis. Am J Obstet Gynecol. 2014 Nov;211(5):453-60. doi: 10.1016/j.ajog.2014.06.014. Epub 2014 Jun 6. PMID 24912096
- [Background] Hesselman S, Hogberg U, Ekholm-Selling K, Rassjo EB, Jonsson M. The risk of uterine rupture is not increased with single- compared with double-layer closure: a Swedish cohort study. BJOG. 2015 Oct;122(11):1535-41. doi: 10.1111/1471-0528.13015. Epub 2014 Aug 4. PMID 25088680
- [Background] Clark EA, Silver RM. Long-term maternal morbidity associated with repeat cesarean delivery. Am J Obstet Gynecol. 2011 Dec;205(6 Suppl):S2-10. doi: 10.1016/j.ajog.2011.09.028. Epub 2011 Oct 6. PMID 22114995
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581
- [Background] Bij de Vaate AJ, van der Voet LF, Naji O, Witmer M, Veersema S, Brolmann HA, Bourne T, Huirne JA. Prevalence, potential risk factors for development and symptoms related to the presence of uterine niches following Cesarean section: systematic review. Ultrasound Obstet Gynecol. 2014 Apr;43(4):372-82. doi: 10.1002/uog.13199. PMID 23996650
- [Background] Dodd JM, Anderson ER, Gates S, Grivell RM. Surgical techniques for uterine incision and uterine closure at the time of caesarean section. Cochrane Database Syst Rev. 2014 Jul 22;2014(7):CD004732. doi: 10.1002/14651858.CD004732.pub3. PMID 25048608
- [Background] Di Spiezio Sardo A, Saccone G, McCurdy R, Bujold E, Bifulco G, Berghella V. Risk of Cesarean scar defect following single- vs double-layer uterine closure: systematic review and meta-analysis of randomized controlled trials. Ultrasound Obstet Gynecol. 2017 Nov;50(5):578-583. doi: 10.1002/uog.17401. Epub 2017 Oct 9. PMID 28070914
- [Background] Hanacek J, Vojtech J, Urbankova I, Krcmar M, Krepelka P, Feyereisl J, Krofta L. Ultrasound cesarean scar assessment one year postpartum in relation to one- or two-layer uterine suture closure. Acta Obstet Gynecol Scand. 2020 Jan;99(1):69-78. doi: 10.1111/aogs.13714. Epub 2019 Sep 26. PMID 31441500
- [Background] Stegwee SI, Jordans IPM, van der Voet LF, Bongers MY, de Groot CJM, Lambalk CB, de Leeuw RA, Hehenkamp WJK, van de Ven PM, Bosmans JE, Pajkrt E, Bakkum EA, Radder CM, Hemelaar M, van Baal WM, Visser H, van Laar JOEH, van Vliet HAAM, Rijnders RJP, Sueters M, Janssen CAH, Hermes W, Feitsma AH, Kapiteijn K, Scheepers HCJ, Langenveld J, de Boer K, Coppus SFPJ, Schippers DH, Oei ALM, Kaplan M, Papatsonis DNM, de Vleeschouwer LHM, van Beek E, Bekker MN, Huisjes AJM, Meijer WJ, Deurloo KL, Boormans EMA, van Eijndhoven HWF, Huirne JAF. Single- versus double-layer closure of the caesarean (uterine) scar in the prevention of gynaecological symptoms in relation to niche development - the 2Close study: a multicentre randomised controlled trial. BMC Pregnancy Childbirth. 2019 Mar 4;19(1):85. doi: 10.1186/s12884-019-2221-y. PMID 30832681
- [Background] Dahlke JD, Mendez-Figueroa H, Maggio L, Sperling JD, Chauhan SP, Rouse DJ. The Case for Standardizing Cesarean Delivery Technique: Seeing the Forest for the Trees. Obstet Gynecol. 2020 Nov;136(5):972-980. doi: 10.1097/AOG.0000000000004120. PMID 33030865